CLINICAL TRIAL: NCT00783289
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety and Tolerability of Multiple-dose Subcutaneous Administration of MEDI-563, a Humanized Anti-interleukin-5 Receptor Alpha Monoclonal Antibody, in Adults With Asthma
Brief Title: A Phase 2a Study to Evaluate the Safety and Tolerability of Benralizumab (MEDI-563) in Adults With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP197
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Asthma
Keywords: Asthma; Benralizumab; MEDI-563
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo matched to benralizumab (MEDI-563) injection subcutaneously on Day 0, 28, and 56.
  Interventions: Other: Placebo
- Benralizumab 25 mg (Experimental): Benralizumab (MEDI-563) injection 25 milligram (mg) subcutaneously on Day 0, 28, and 56.
  Interventions: Biological: Benralizumab 25 mg
- Benralizumab 100 mg (Experimental): Benralizumab (MEDI-563) injection 100 mg subcutaneously on Day 0, 28, and 56.
  Interventions: Biological: Benralizumab 100 mg
- Benralizumab 200 mg (Experimental): Benralizumab (MEDI-563) injection 200 mg subcutaneously on Day 0, 28, and 56.
  Interventions: Biological: Benralizumab 200 mg

INTERVENTIONS:
Other: Placebo — Placebo matched to benralizumab (MEDI-563) injection subcutaneously on Day 0, 28, and 56.
  Arms: Placebo
Biological: Benralizumab 25 mg — Benralizumab (MEDI-563) injection 25 milligram (mg) subcutaneously on Day 0, 28, and 56.
  Other Names: MEDI-563
  Arms: Benralizumab 25 mg
Biological: Benralizumab 100 mg — Benralizumab (MEDI-563) injection 100 mg subcutaneously on Day 0, 28, and 56.
  Other Names: MEDI-563
  Arms: Benralizumab 100 mg
Biological: Benralizumab 200 mg — Benralizumab (MEDI-563) injection 200 mg subcutaneously on Day 0, 28, and 56.
  Other Names: MEDI-563
  Arms: Benralizumab 200 mg

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of escalating multiple subcutaneous (SC) doses of MEDI-563 in adult subjects with asthma.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, dose-escalation, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of multiple subcutaneous doses (25, 100, or 200 milligram [mg]) of benralizumab (MEDI-563) in adult subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Age 18 through 80 years at screening
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Previously documented diagnosis of asthma of more than or equal to (>=) 1 year duration, based on episodic symptoms of airflow obstruction; post-bronchodilator reversibility of airflow obstruction >=12 percent (%) (at screening or documented within 1 year prior to randomization); or proof of a positive response to a methacholine challenge (documented within 1 year prior to randomization) as represented by a provoking concentration of methacholine to cause a 20% fall in forced expiratory volume in 1 second (FEV1); (PC20) less than (<) 8 milligram per milliliter (mg/mL)
* Weight of >=45 kilogram (kg) but less than or equal to (<=) 135 kg (>=100 pounds [lb] but <=300 lb)
* Able to produce spirometry readings that meet American Thoracic Society (ATS)/European Respiratory Society (ERS) standards
* Screening pre-bronchodilator FEV1 >=60%
* Women of childbearing potential, unless surgically sterile (including tubal ligation) and/or at least 2 years post-menopausal, must use 2 effective methods of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of a condom with spermicide by the sexual partner, or sterile sexual partner) for 14 days prior to the first dose of the investigational product on Study Day 0, and must agree to continue using such precautions through Study Day 161. Cessation of birth control after this point should be discussed with a responsible physician
* Men, unless surgically sterile, must likewise use 2 effective methods of birth control (for example, condom with spermicide) and must agree to continue using such contraceptive precautions through End of Study/Study Day 161
* Ability to complete the study period, including follow-up period until Study Day 161 as required by protocol

Exclusion Criteria:

* Previously received benralizumab (MEDI-563)
* History of allergy or reaction to any component of the investigational product formulation
* History of allergy or reaction to any other marketed or experimental monoclonal antibody therapies, intravenous gammaglobulin (IVIG), or blood products
* Receipt of any investigational drug therapy within 30 days prior to randomization into the study or any biologic(s) within 5 half-lives of the agent prior to randomization into the study
* Treatment with an oral or systemic burst of corticosteroids within 4 weeks prior to randomization into the study
* Use of any chronic systemic immunosuppressive drugs, including oral corticosteroids within 4 weeks prior to randomization into the study
* Current use of any oral or ophthalmic beta-adrenergic antagonist (for example, propranolol), must have been stopped 2 weeks prior to randomization into the study
* Current allergy vaccination (immunotherapy)
* History of anaphylaxis
* Lung disease other than persistent asthma (for example, chronic bronchitis, cystic fibrosis, chronic obstructive pulmonary disease [COPD], tuberculosis [TB])
* Acute illnesses or evidence of significant active infection, such as fever >=38.0 degrees Celsius [C] (>=100.5 degrees Fahrenheit [F]) at screening and up through time of the first dose of the investigational product
* History of ingestion of untreated water in a location known to be infected with parasites, resulting in acute or chronic diarrhea; or an untreated parasitic infection within 1 month of randomization
* Pregnancy (women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to administration of the investigational product)
* Lactating woman
* Infection with human immunodeficiency virus (HIV)-1, HIV-2, or hepatitis A, B, or C virus
* History of cancer, apart from basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy >= 1 year prior to randomization into the study
* History of cigarette smoking >=10 pack years
* History of alcohol abuse or drug abuse that required treatment <1 year prior to randomization into the study
* Elective surgery planned during the study period
* Evidence of any systemic disease or any finding upon physical examination, laboratory abnormality, chest x-ray (CXR), or electrocardiogram (ECG) that, in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or confound the analysis of the study results
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or first degree family members of such individuals (that is, parents, siblings, or children)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11-14 (Actual); Primary Completion 2009-11-17 (Actual); Study Completion 2009-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gossage, M.D., Study Director — MedImmune LLC
Locations (6):
- United States (6):
  - Research Site, Encinitas, California
  - Research Site, Los Angeles, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Wheaton, Maryland
  - Allergy Associates Research Center, Portland, Oregon
  - Research Site, Upland, Pennsylvania

REFERENCES:
- See also: Attachments tab: MI-CP197 Redacted Protocol_22_Jul_2015 — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/View?id=64

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Started | 6 | 7 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.2) | 50.4 (12.3) | 45.5 (13.4) | 40.2 (12.5) | 45.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 3 | 14
  Male | 3 | 3 | 2 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Day 161 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 0 to Day 161
Population: Safety population included all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
participants
  TEAEs | 3 | 4 | 4 | 4
  TESAEs | 0 | 0 | 0 | 0

2. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for Benralizumab
Time Frame: Day 0, 1, 7, 28, 35, 56, 84, 112, and 161
Population: Safety population included all participants who received at least 1 dose of the investigational product. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: days
Arm/Group | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Number analyzed (Participants) | 6 | 6 | 6
days | 7.00 [7.00 to 28.00] | 7.00 [1.00 to 7.00] | 7.00 [7.00 to 7.00]

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Benralizumab
Time Frame: Day 0, 1, 7, 28, 35, 56, 84, 112, and 161
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Number analyzed (Participants) | 6 | 6 | 6
microgram per milliliter (mcg/mL) | 1.152 (0.615) [7 to 28] | 4.127 (1.775) [1 to 7] | 15.637 (8.062) [7 to 7]

4. Secondary Outcome: Area Under the Curve From Time 0 to Infinity (AUC [0-infinity]) for Benralizumab
Description: Area under the serum concentration-time curve from time-zero extrapolated to infinity postdose.
Time Frame: Day 0, 1, 7, 28, 35, 56, 84, 112, and 161
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter
Arm/Group | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Number analyzed (Participants) | 4 | 4 | 4
microgram*day per milliliter | 118.335 (69.640) [7 to 28] | 405.868 (205.856) [1 to 7] | 1157.013 (86.444) [7 to 7]

5. Secondary Outcome: Terminal Phase Elimination Half-Life (t1/2) for Benralizumab
Description: Terminal phase elimination half-life (t1/2) is the time measured for the serum concentration to decrease by one half.
Time Frame: Day 0, 1, 7, 28, 35, 56, 84, 112, and 161
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Number analyzed (Participants) | 4 | 4 | 4
days | 17.163 (2.368) [7 to 28] | 18.610 (3.905) [1 to 7] | 18.315 (3.484) [7 to 7]

6. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies (ADAs) to Benralizumab at Any Visit
Time Frame: Day 0, 28, 56, 84, 112, and 161
Population: Safety population included all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
participants | 0 | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: Day 0 to Day 161
Arm/Group | Placebo | Benralizumab 25 mg | Benralizumab 100 mg | Benralizumab 200 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 4/7 | 4/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Benralizumab 25 mg (N=7) | Benralizumab 100 mg (N=6) | Benralizumab 200 mg (N=6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.